CLINICAL TRIAL: NCT03701893
Title: Evaluate the Effect of the Strain Lactobacillus PS11610 on the Microbiota of the Female and Male Genital Tract in Couples With Fertility Problems and Dysbiosis.
Brief Title: Evaluate the Use of a New Probiotic Strain in Couples With Fertility Problems and Dysbiosis.
Acronym: PROFEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FEC/18.01
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Infertility; Vaginal Flora Imbalance; Genital Disorder
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Open label intervention study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactobacillus PS11610 (Experimental): Lactobacillus PS11610 for couples with genital dysbiosis and infertility. Each dose contains 1*10E9 colony forming unit (CFU) of Lactobacillus PS11610.Two daily doses for her and one daily dose for him until pregnancy or end of study period (6 months).
  Interventions: Dietary Supplement: Lactobacillus PS11610

INTERVENTIONS:
Dietary Supplement: Lactobacillus PS11610 — 7 months and a half intervention study. A 6 months intervention period preceded by a period of sampling and analysis of vaginal, seminal and gland swabs of 6 weeks. During the 6 months of intervention the men participants will intake one capsule that contains 1*10E9 colony forming unit (CFU) of Lactobacillus PS11610 and the women participating will intake two capsules of the same product (each 12 hours). If the couple stay pregnant during the intervention the man will end the product intake and the woman will reduce the dose to one capsule with 1*10E9 CFU of Lactobacillus PS11610 per day during 12 additional weeks.

SUMMARY:
Pilot study to evaluate the effect of the strain Lactobacillus PS11610 on the microbiota of the female and male genital tract in couples with fertility problems. Couples who have started treatment for artificial insemination or who are on the waiting list for an invitro fertilization treatment will be invited to participate. The estimated duration of the study will be 7 and a half months.

DETAILED DESCRIPTION:
Pilot study to evaluate the effect of the strain Lactobacillus PS11610 on the microbiota of the female and male genital tract in couples with fertility problems. Couples who have started treatment for artificial insemination or who are on the waiting list for an invitro fertilization treatment will be invited to participate. The estimated duration of the study will be 7 and a half months.

Four visits are included in the study period.

ELIGIBILITY:
Inclusion Criteria:

* Couples with ages between 20 and 40
* Couples under an assisted reproduction treatment: Artificial Insemination or In vitro Fertilization.
* Signature of informed consent

Exclusion Criteria:

* Anovulation
* Hyperprolactinemia
* Hypogonadotropic hypergonadism
* Hypergonadotropic Hypergonadism
* Hyperandrogenisms
* Polycystic ovary syndrome
* Endometriosis
* Pelvic adhesions
* Myomas, polyps and / or uterine synechia
* Diagnosis of tubal factor (hydrosalpinx, tubal obstructions)
* Low ovarian reserve
* Azoospermia
* Sperm motility (A + B) <25%
* Sperm morphology ≤2%
* With chronic diseases that cause intestinal malabsorption
* With known congenital or acquired immunodeficiency.
* Obesity (IMC ≥ 30)
* Current history or diagnosis of alcohol, tobacco and drug abuse
* Uncertainty about the willingness or ability of the participants to comply with the requirements of the protocol.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Counts of microorganisms presents in cultured samples of genital tracts obtained from infertility couples. | 7 months and a half
  The microbial composition obtained by culture of genital tracts samples from couples with infertility

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manzano, PhD, Study Chair — ProbiSearch SL
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided